CLINICAL TRIAL: NCT05076812
Title: Interleukin 38 as a Biomarker for Metabolic Syndrome in Psoriatic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yomna Abdo Abdellatif, resident doctor in dermatology venereology and andrology department in sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-09-02
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Psoriasis
Keywords: psoriasis; metabolic syndrome; interleukin 38
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (4):
- Group 1 (Psoriasis only): contains 24 psoriatic patients, Psoriasis Area Severity Index will be measured, also waist circumference, body mass index, blood pressure, fasting blood glucose and fasting lipid profile and finally: plasma level of interleukin 38
  Interventions: Diagnostic Test: measure plasma level of interleukin 38 by ELISA kit
- Group 2 (Psoriasis and metabolic syndrome): contains 24 psoriatic patients with metabolic syndrome. Psoriasis Area Severity Index will be measured metabolic syndrome is diagnosed after measuring waist circumference, body mass index, blood pressure, fasting blood glucose and fasting lipid profile finally: plasma level of interleukin 38
  Interventions: Diagnostic Test: measure plasma level of interleukin 38 by ELISA kit
- Group 3 (Metabolic syndrome only): contains 24 patients with metabolic syndrome only. full dermatological examination to exclude psoriasis and other inflammatory skin disorders metabolic syndrome is diagnosed after measuring waist circumference, body mass index, blood pressure, fasting blood glucose and fasting lipid profile finally: plasma level of interleukin 38
  Interventions: Diagnostic Test: measure plasma level of interleukin 38 by ELISA kit
- Group 4 (Healthy Controls): contains 24 healthy control subjects full dermatological examination to exclude psoriasis and other inflammatory skin disorders metabolic syndrome is excluded after measuring waist circumference, body mass index, blood pressure, fasting blood glucose and fasting lipid profile finally: plasma level of interleukin 38
  Interventions: Diagnostic Test: measure plasma level of interleukin 38 by ELISA kit

INTERVENTIONS:
Diagnostic Test: measure plasma level of interleukin 38 by ELISA kit — draw 5 ml of venous blood into EDTA tubes and centrifuged then plasma is separated for test

SUMMARY:
case control study to compare level of interleukin 38 in patients with psoriasis and patients with metabolic syndrome with healthy control subjects

DETAILED DESCRIPTION:
this case control study will measure plasma level of interleukin 38 in 4 groups of 24 subject, group one will have psoriatic patients, group 2 will have psoriatic patients with metabolic syndrome, group three will have patients with metabolic syndrome only, and group 4 will have healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* specific to each group

Exclusion Criteria:

* Patient refusal. Age <18 years Pregnancy Lactation smoking Infections. Patients with other inflammatory skin disorders use of antioxidant and anti-inflammatory drugs patients on treatment for psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people attending the Dermatology Outpatient Clinics of Sohag University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
measure plasma level of interleukin 38 in all groups | through study completion an average of 18 months
  level of interleukin 38 will be measured and compared in all groups to asses the relationship between this interleukin and metabolic syndrome in psoriatic patients

CONTACTS AND LOCATIONS:
Overall Officials: yomna a abdellatif, MBBCH, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided